CLINICAL TRIAL: NCT02508090
Title: Long-Term Extension to a Phase 2, Open-Label, Clinical Trial of Miravirsen Sodium in Null Responders to Pegylated-Interferon Alpha Plus Ribavirin in Subjects With Chronic Hepatitis C (CHC) Virus Genotype 1 Infection
Brief Title: Long-Term Extension Study of Miravirsen Among Participants With Genotype 1 Chronic Hepatitis C (CHC) Who Have Not Responded to Pegylated-Interferon Alpha Plus Ribavirin
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Santaris Pharma A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NP29711; NCT02031133 (obsolete NCT alias)
Record Dates: First submitted 2015-07-23; First posted 2015-07-24 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine samples will be collected over a course of 7 study visits to obtain hematology, chemistry, urinalysis, coagulation, HCV RNA, and viral resistance data.

GROUPS / COHORTS (1):
- Study Population: Participants who previously received 12 weeks of miravirsen monotherapy in Study SPC3649-207 will complete up to 36 months of safety and efficacy follow-up without investigational treatment.

SUMMARY:
Genotype 1 CHC participants from Study SPC3649-207 with null response to prior pegylated-interferon alpha plus ribavirin will be enrolled into this 36-month extension study, designed to evaluate the long-term safety and efficacy after 12 weeks of miravirsen monotherapy. Due to the observational nature of the study, miravirsen will not be dosed as an investigational product.

ELIGIBILITY:
Inclusion Criteria:

* Participants from Study SPC3649-207, including those who completed the study and those who discontinued or terminated the study early for any reason, or those who opted to receive other approved therapy for the treatment of hepatitis C virus (HCV) infection

Exclusion Criteria:

* Participants who have received investigational drug therapy after discontinuation, termination, or completion of Study SPC3649-207

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will enroll null responders with CHC genotype 1 virus infection who have participated in Study SPC3649-207.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-08-02 (Actual); Primary Completion 2017-01-13 (Actual); Study Completion 2017-01-13 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 36 months
Incidence of sustained virologic response (SVR) | 48 weeks after end of treatment (EOT)
Change from Baseline in HCV ribonucleic acid (RNA) level | Up to 36 months
Incidence of HCV resistance | Up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Fundacion de Investigacion de Diego, San Juan, Puerto Rico